CLINICAL TRIAL: NCT04596111
Title: Can Aerobic and Anaerobic Fitness Tests be Used to Track Rowing Performance Changes in Collegiate Rowers?
Brief Title: Physiological Variables and Rowing Performance.
Status: Completed | Type: Observational
Sponsor: Franklin Pierce University (Other)
Responsible Party: Principal Investigator, Tongyu Ma, Assistant Professor of Health Sciences, Franklin Pierce University
Other Study IDs: YB09042020
Record Dates: First submitted 2020-10-11; First posted 2020-10-22 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Water Sports

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to investigate the association between the changes in physiological variables based on fitness testing and the changes in rowing performance.

DETAILED DESCRIPTION:
The literature has shown that both aerobic capacity and anaerobic capacity are important for exercise performance in rowing. Simple fitness tests (e.g., the modified Wingate test and the graded exercise test) have been validated to examine aerobic and anaerobic capacities in rowers. However, it remains unclear whether these fitness tests can be used to track rowing performance changes. The purpose of this study is to investigate the association between the changes in fitness test outcomes and the changes in rowing performance. The investigators expect that improvements in rowing performance are closely related to improvements in fitness test outcomes.

Participants will attend two sessions of fitness testing, one in the fall 2020 and one in the spring 2021. Each session will include the modified Wingate test to examine anaerobic capacity, the graded exercise test to examine the aerobic capacity, and the 2,000-meter rowing test on rowing ergometers to assess rowing performance.

Modified Wingate test:

After 3 minutes of warm-up at 40-50% of heart rate reserve, the participants will perform 30 seconds of rowing at maximal effort on the rowing ergometer.

Graded exercise test:

Workload will start from 25 Watts and it will be increased by 25 Watts by each stage until exhaustion. Each stage includes 2 minutes of rowing and 1 minute of rest.

2,000-meter rowing test: A 2,000-meter race simulation will be performed using an indoor rowing ergometer.

ELIGIBILITY:
Inclusion Criteria:

• Collegiate rowers

Exclusion Criteria:

* Cardiovascular diseases
* Pulmonary diseases
* Metabolic diseases
* Other contraindications to exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be current rowers of a college rowing team.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Rowing performance | six months
  Time to complete the 2,000-meter indoor rowing test

SECONDARY OUTCOMES:
Maximal oxygen consumption | six months
  The highest oxygen consumption during a graded exercise test.
Maximal anaerobic power | six months
  The maximal power output during a 30-second anaerobic test.

CONTACTS AND LOCATIONS:
Overall Officials: Tongyu Ma, Ph.D., Study Director — Franklin Pierce University
Locations (1):
- Franklin Pierce University, Rindge, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No